CLINICAL TRIAL: NCT06382961
Title: Postoperative Infusion of Dexmedetomidine for Prevention of Postoperative Delirium in Elderly Patients Undergoing Lung Surgery: A Randomized Controlled Trial
Brief Title: Postoperative Dexmedetomidine in Prevention of Postoperative Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Intelligent Medical Research Center, Shenzhen United Scheme Technology Co., Ltd. (Industry)
Collaborators: Shenzhen People's Hospital (Other); Dongyuan People's Hospital (Unknown); Kunming Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SZUS_231101
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Delirium in Old Age; Anesthesia; Adverse Effect
MeSH Terms: interventions — Dexmedetomidine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental)
  Interventions: Drug: Dexmedetomidine injection
- Control (Active Comparator)
  Interventions: Drug: Sufentanil injection

INTERVENTIONS:
Drug: Dexmedetomidine injection — Combining with 3 μg.kg-1 sufentanil, 3 μg.kg-1 dexmedetomidine is injected through intravenous patient controlled anesthesia pump in a 2 ml bolus with 20 minutes lock-out, and a background infusion rate of 2 ml per hour.
  Arms: Experiment
Drug: Sufentanil injection — 3 μg.kg-1 sufentanil is injected through intravenous patient controlled anesthesia pump in a 2 ml bolus with 20 minutes lock-out, and a background infusion rate of 2 ml per hour.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn how postoperative infusion of dexmedetomidine would influence postoperative delirium in elderly patients undergoing lung surgery. The main questions it aims to answer are :

1. Does postoperative dexmedetomidine reduce the incidence of delirium after lung surgery?
2. Does postoperative dexmedetomidine introduce other medical problems? Researchers will compare dexmedetomidine and sufentanil to see if dexmedetomidine works to reduce delirium.

Participants will undergo routine postoperative care:

1. Patient-controlled self anesthesia with sufentanil only or combination of sufentanil and dexmedetomidine
2. Postoperative visit twice a day for at least seven days

ELIGIBILITY:
Inclusion Criteria:

* elective surgery for lobectomy or segmentectomy

Exclusion Criteria:

* local allergy to anesthetics;
* patients with a clear preoperative history of nervous system and mental system diseases or long-term use of sedatives or antidepressants;
* history of alcoholism, drug abuse or drug dependence;
* have a history of brain surgery or injury;
* epilepsy and associated mental and cognitive dysfunction, long-term stress stimulation, or psychological disorders;
* sick sinus syndrome, second-degree or greater atrioventricular block or other contraindications for use of α2 adrenergic agonist;
* liver and kidney insufficiency.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 287 (Actual)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Delirium is assessed at 8 am and 8 pm for 3 days after surgery

SECONDARY OUTCOMES:
Incidence of postoperative nausea and vomiting | Assessed twice a day for 7days after surgery
incidence of postoperative complications | Assessed daily for 3 days after surgery
  Other postoperative complications including including hypotension, hypertension, bradycardia, tachycardia, and hypoxemia
Pain intensities | Assessed daily at 8 am for 3 days after surgery
  patient pain assessed using numeric rating scale, ranged from 0 to 11, higher score indicate higher pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Rui Zhao, Study Director — Department of Anesthesiology, Kunming Children's Hospital
Locations (1):
- Kunming Children's Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No